CLINICAL TRIAL: NCT00578448
Title: An Open-label Pharmacokinetic Study in De Novo Renal Transplant Subjects Receiving a Belatacept Based Immunosuppressant Regimen
Brief Title: Belatacept Pharmacokinetic Trial in Renal Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM103-047
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): 10mg/kg
  6 doses (Day 1, 5, week 2, 4, 8 and 12) for 12 weeks
  Interventions: Drug: Belatacept
- B (Active Comparator): 5mg/kg
  33 doses (every 4 weeks) for 144 weeks
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — IV infusion
  Other Names: BMS-224818

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of belatacept in de novo renal transplant subjects treated with belatacept-based immunosuppressant medication

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a living or deceased donor kidney
* First or second transplant
* Men and women, including women of childbearing potential, 18 years and older

Exclusion Criteria:

* Panel reactive antibodies ≥ 30%
* Significant infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (2):
  - Western New England Renal & Transplant, Springfield, Massachusetts
  - Henry Ford Hospital, Detriot, Michigan
- Local Institution, Capital Federal, Buenos Aires, Argentina
- Mexico (2):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Cuernavaca, Morelos

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant, first visit: 3 March 2008. Last subject, last visit 6 September 2012. Participants had received a renal transplant from a living or deceased donor with an anticipated cold ischemia time of less than (<) 24 hours (h)
Pre-assignment Details: 14 participants enrolled; 12 received study drug; 2 not treated due to: kidney damage (1) and prolonged cold ischemia (1). Study continued for up to 3 years until drug approval in participant's country. Participants continued in a 1 year extension after conclusion of the 3rd year.
Groups:
- Belatacept 10mg/kg; 5mg/kg Maintenance: Participants received intravenous (IV) belatacept (10 milligram per kilogram body weight (mg/kg) on Days 1 and 5, and then every 2 weeks through Month 1 (Weeks 2 and 4), and then every 4 weeks through Month 4 (Weeks 8 and 12). After 4 months, participants received a maintenance dose of 5 mg/kg belatacept administered every 4 weeks until completion of the trial (3 years and then a 1 year extension was available for those who completed the 3rd year).
Period: Day 1 up to 3 Years of Planned Study
Arm/Group | Belatacept 10mg/kg; 5mg/kg Maintenance
Started | 12
Completed | 9
Not Completed | 3
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — started marketed Cellcept and Prograf | 1
Period: 1 Year Long Term Extension (LTE)
Arm/Group | Belatacept 10mg/kg; 5mg/kg Maintenance
Started | 9
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Participants treated with study drug after renal transplant.
Groups:
- IV Belatacept 10mg/kg With 5mg/kg Maintenance: Participants received intravenous (IV) belatacept (10 milligram per kilogram body weight (mg/kg) on Days 1 and 5, and then every 2 weeks through Month 1 (Weeks 2 and 4), and then every 4 weeks through Month 4 (Weeks 8 and 12). After 4 months, participants received a maintenance dose of 5 mg/kg belatacept administered every 4 weeks until completion of the trial.
Arm/Group | IV Belatacept 10mg/kg With 5mg/kg Maintenance
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (19.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 4
  Mexico | 6
  Argentina | 2
Weight [Mean (Standard Deviation); unit: kilograms] | 74.90 (17.735)

OUTCOME MEASURES:

1. Primary Outcome: Mean Belatacept Serum Concentrations Between Weeks 12 and 16 by Nominal Collection Time, Following 10mg/kg IV Belatacept - Pharmacokinetic Population
Description: Pharmacokinetic (PK) sampling started from pre-dose (0 hour) on Day 84 and ended at 672 hour (h) on Day 112 (between Weeks 12 to 16). The samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method and measured as nanograms/milliliter (ng/mL). Less than the lower limit of quantification (LLQ), 3.000 ng/mL concentration value was treated as missing.
Time Frame: Day 84 to Day 112
Population: Number (N) of participants analyzed for each collection time was 10, except for time 0.50 h, which was missing 1 participant. Therefore Number (N) for Time 0.50 h = 9.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance: Participants received intravenous (IV) belatacept (10 milligram per kilogram body weight (mg/kg) on Days 1 and 5, and then every 2 weeks through Month 1 (Weeks 2 and 4), and then every 4 weeks through Month 3. After Day 112, participants received a maintenance dose of 5 mg/kg belatacept administered every 4 weeks until completion of the study.
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 10
ng/mL
  0.00 h | 8491.00 (5175.97)
  0.50 h | 242667 (64459.3)
  2.00 h | 212800 (62467.4)
  72.00 h | 55970.0 (12989.7)
  168.00 h | 36890.0 (16426.8)
  336.00 h | 19063.0 (7803.41)
  504.00 h | 11587.0 (6282.26)
  672 h | 7613.00 (4698.61)

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) Between Weeks 12 and 16 Following 10mg/kg IV Belatacept and Trough Serum Concentration Prior to Dosing (Cmin) - Pharmacokinetic Population
Description: Cmax, Cmin are measured in micrograms per milliliter (µg/mL). At Day 84, blood samples obtained from pre-dose (0 hour) and ended at 672 hour (h) on Day 112. Serum samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method. Individual participant PK parameters were derived from serum concentration versus time data using a non-compartmental method, using a validated PK analysis program (KineticaTM 4.4.1 within the eToolbox [version 2.6.1]). Actual sampling times were used for PK calculations. The Cmax, and the Cmin were recorded directly from experimental observations. Using no weighting factor, the terminal log-linear phase of the concentration-time curve was identified by least-square linear regression of at least 3 data points that yielded a maximum G-criteria, which is also referred to as adjusted R-squared. Values below lower limits of quantification (LLQ), 0.003 µg/mL, were set to 0.0015 for computation of summary statistics.
Time Frame: Day 84 to Day 112
Population: One participant excluded from analysis of Cmax and Tmax due to a very high concentration value (it was considered an outlier) therefore, for Cmax, Number of participants analyzed (N)=9.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 10
µg/mL
  Cmin | 7.29 (61)
  Cmax | 238.33 (27)

3. Primary Outcome: Time of Maximum Observed Serum Concentration (Tmax) Between Weeks 12 and 16 Following 10mg/kg IV Belatacept - Pharmacokinetic Population
Description: Tmax measured in hours (h). At Day 84, blood samples obtained from pre-dose (0 hour) and ended at 672 (h) on Day 112 . The samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method. Individual participant PK parameters were derived from serum concentration versus time data using a non-compartmental method, using a validated PK analysis program (KineticaTM 4.4.1 within the eToolbox [version 2.6.1]). Actual sampling times were used for PK calculations.
Time Frame: Day 84 to Day 112
Population: 1 participant excluded from analysis of Cmax and Tmax due to a very high concentration value (it was considered an outlier) therefore, for Tmax, Number of participants analyzed (N)=9.
Measure: Median (Full Range); unit: hours
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 9
hours | 0.60 [0.5 to 2.5]

4. Primary Outcome: Area Under the Concentration Time Curve Within a Dosing Interval (AUC) (TAU) Between Weeks 12 and 16 Following 10 mg/kg IV Belatacept - Pharmacokinetic Population
Description: At Day 84, blood samples obtained from pre-dose (0 hour) and ended at 672 hour (h) on Day 112. The samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method. Individual participant PK parameters were derived from serum concentration versus time data using a non-compartmental method, using a validated PK analysis program (KineticaTM 4.4.1 within the eToolbox [version 2.6.1]). The area under the concentration-time curve in one dose interval [AUC(TAU), where TAU = 4 weeks] were calculated using the mixed log-linear trapezoidal algorithm in Kinetica. Actual sampling times were used for PK calculations. AUC (TAU) was measured as micrograms multiplied by time(h) per milliliter (µg*h/mL).
Time Frame: Day 82 to Day 112
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 10
µg*h/mL | 21241 (35)

5. Secondary Outcome: Summary of Trough Serum Concentration of Belatacept Prior to Dosing up to 3 Years Post Transplantation - Pharmacokinetic Population
Description: Blood samples were obtained pre and post dose at designated time points up to Day 112 and thereafter, pre-dose samples were obtained at Days 168 and 364, and then once yearly up to end of Year 3. The samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method. Individual participant PK parameters were derived from serum concentration versus time data using a non-compartmental method, using a validated PK analysis program (KineticaTM 4.4.1 within the eToolbox [version 2.6.1]). Actual sampling times were used for PK calculations. The trough serum concentration (Cmin), was recorded directly from experimental observations. Using no weighting factor, the terminal log-linear phase of the concentration-time curve was identified by least-square linear regression of at least 3 data points that yielded a maximum G-criteria, which is also referred to as adjusted R-squared. Cmin was measured as micrograms per milliliter (µg/mL).
Time Frame: Day 1 to Day 1092
Population: Number of participants (N) analyzed = 11 for Days 5, 14,and 28; and 12 for Day 56. Days 84, 112, 168, 364 N=10.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- 10mg/kg IV Belatacept: Participants received intravenous (IV) belatacept (10 milligram per kilogram body weight (mg/kg) on Days 1 and 5, and then every 2 weeks through Month 1 (Weeks 2 and 4), and then every 4 weeks through Month 3. After Day 112, participants received a maintenance dose of 5 mg/kg belatacept administered every 4 weeks until completion of the study.
Arm/Group | 10mg/kg IV Belatacept
Number analyzed (Participants) | 11
µg/mL
  Day 5 Post Transplantation | 33.499 (25.020)
  Day 14 Post Transplantation | 24.558 (40.605)
  Day 28 Post Transplantation | 21.375 (39.224)
  Day 56 Post Transplantation (N=12) | 8.574 (58.386)
  Day 84 Post Transplantation | 7.289 (60.959)
  Day 112 Post Transplantation | 6.391 (61.718)
  Day 168 Post Transplantation | 3.189 (47.797)
  Day 364 Post Transplantation | 3.704 (42.236)
  Day 728 Post Transplantation | 4.383 (43.209)
  Day 1092 Post Transplantation | 4.996 (55.892)

6. Primary Outcome: Total Body Clearance (CLT) Between Weeks 12 and 16 Following 10mg/kg IV Belatacept - Pharmacokinetic Population
Description: At Day 84, blood samples obtained from pre-dose (0 hour) and ended at 672 hour (h) on Day 112. The samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method. Individual participant PK parameters were derived from serum concentration versus time data using a non-compartmental method, using a validated PK analysis program (KineticaTM 4.4.1 within the eToolbox [version 2.6.1]). Actual sampling times were used for PK calculations. CLT was calculated by dividing the dose by AUC(TAU) and was adjusted to body weight. CLT was measured as milliliter per time per kg body weight (mL/h/kg).
Time Frame: Day 84 to Day 112
Population: Participants who were treated and had PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 10
mL/h/kg | 0.47 (27)

7. Primary Outcome: Steady-state Volume Distribution (Vss) Following 10mg/kg IV Belatacept Between Weeks 12 and 16 - Pharmacokinetic Population
Description: At Day 84, blood samples obtained from pre-dose (0 hour) and ended at 672 hour (h) on Day 112. The samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method. Individual participant PK parameters were derived from serum concentration versus time data using a non-compartmental method, using a validated PK analysis program (KineticaTM 4.4.1 within the eToolbox [version 2.6.1]). Actual sampling times were used for PK calculations. Vss was calculated by dividing the dose by AUC and multiply the mean residence time (MRT). Vss was adjusted to body weight and measured as liter per kilogram body weight (l/kg).
Time Frame: Day 84 to Day 112
Measure: Mean (Standard Deviation); unit: l/kg
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 10
l/kg | 0.11 (0.033)

8. Primary Outcome: Serum Half Life (T-HALF) Between Weeks 12 and 16 Following 10mg/kg IV Belatacept - Pharmacokinetic Population
Description: At Day 84, blood samples obtained from pre-dose (0 hour) and ended at 672 hour (h) on Day 112. The samples were analyzed for belatacept by enzyme-linked immunosorbent assay (ELISA) using a validated method. Individual participant PK parameters were derived from serum concentration versus time data using a non-compartmental method, using a validated PK analysis program (KineticaTM 4.4.1 within the eToolbox [version 2.6.1]). Actual sampling times were used for PK calculations. T-HALF was calculated as ln2/Lz, where Lz is the absolute value of the slope of the terminal log-linear phase. T-HALF is measured in hours (h).
Time Frame: Day 84 to Day 112
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 10
hours | 235.43 (76.414)

9. Secondary Outcome: Acute Rejection, Graft Loss, and Death up to 3 Years Post Transplantation in Planned Study and 1 Year Long Term Extension - All Treated Participants
Description: Acute rejection of transplant defined as a clinicopathological event requiring clinical evidence and biopsy confirmation by central pathologist. Graft loss was defined as either functional loss or physical loss. Day 1 is day of transplantation.
Time Frame: Day 1 up to 4 years post transplantation
Population: All treated participants were analyzed during the planned 3 year study N=12. Only 9 participants entered the LTE so N=9 for LTE.
Measure: Number; unit: participants
Groups:
- Belatacept 10mg/kg; 5mg/kg Maintenance: Participants received intravenous (IV) belatacept (10 milligram per kilogram body weight (mg/kg) on Days 1 and 5, and then every 2 weeks through Month 1 (Weeks 2 and 4), and then every 4 weeks through Month 3. After Day 112, participants received a maintenance dose of 5 mg/kg belatacept administered every 4 weeks until completion of the study (3 years planned study; 1 year extension allowed to those who completed 3rd year).
Arm/Group | Belatacept 10mg/kg; 5mg/kg Maintenance
Number analyzed (Participants) | 12
participants
  Acute rejection of transplant | 4
  Death | 1
  Graft Loss | 1

10. Secondary Outcome: Mean Change From Baseline to Days 5, 28, 112, 168, and 364 in Tryptophan - All Treated Participants
Description: Indoleamine 2,3 dioxygenase (IDO) is a tryptophan catabolizing enzyme that can be induced in antigen-presenting cells by the engagement of B7 by cytotoxic lymphocyte antigen 4 (CTLA-4). Tryptophan depletion in cellular microenvironments has an inhibitory effect on T cells and may be part of a broader immuno-regulatory effect of IDO induction. The IDO activity was determined by measuring the quantity of tryptophan and its metabolite, kynurenine, in serum samples using a validated high performance liquid chromatography (HPLC) method. Baseline is defined as pre-dose. Tryptophan was measured in micromoles (µM)
Time Frame: Baseline to Day 364
Population: Number analyzed for Baseline, Days 5, 28, 112, 168, 364 = 12, 11, 11, 10, 10, and 10, respectively.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 12
µM
  Day 5 Post Transplantation | -27.375 (38.9151)
  Day 28 Post Transplantation | -22.765 (39.0174)
  Day 112 Post Transplantation | -27.331 (39.2819)
  Day 168 Post Transplantation | -18.627 (37.9010)
  Day 364 Post Transplantation | -24.610 (41.4859)

11. Secondary Outcome: Mean Change From Baseline to Days 5, 28, 112, 168, and 364 in Kynurenine - All Treated Participants
Description: Indoleamine 2,3 dioxygenase (IDO) is a tryptophan catabolizing enzyme that can be induced in antigen-presenting cells by the engagement of B7 by CTLA-4. Tryptophan depletion in cellular microenvironments has an inhibitory effect on T cells and may be part of a broader immuno-regulatory effect of IDO induction. The IDO activity was determined by measuring the quantity of tryptophan and its metabolite, kynurenine, in serum samples using a validated high performance liquid chromatography (HPLC) method. Baseline is defined as pre-dose. Kynurenine was measured in micromoles (µM).
Time Frame: Day 1 to Day 364
Population: Number analyzed for Baseline, Days 5, 28, 112, 168, 364 = 12, 11, 11, 10, 10, and 10, respectively.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Belatacept 10mg/kg(3 Months); 5mg/kg Maintenance
Number analyzed (Participants) | 12
µM
  Day 5 Post Transplantation | -7.276 (9.3070)
  Day 28 Post Transplantation | -8.486 (9.1880)
  Day 112 Post Transplantation | -7.936 (9.6630)
  Day 168 Post Transplantation | -7.589 (9.6115)
  Day 364 Post Transplantation | -7.279 (9.7117)

ADVERSE EVENTS:
Time Frame: Day 1 (day of transplant) up to 3 years post transplant for the study and 1 additional year for the 1 year extension for those participants who entered the extension.
Arm/Group | Bela 10-5mg/kg
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bela 10-5mg/kg (N=12)
Myelopathy (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Pyrexia (General disorders) | 1
Ureteral necrosis (Renal and urinary disorders) | 1
Blood creatine increased (Investigations) | 1
Cellulitis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Meningitis viral (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bela 10-5mg/kg (N=12)
Aneurysm (Vascular disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Eye pain (Eye disorders) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypothyroidism (Endocrine disorders) | 1
Insomnia (Psychiatric disorders) | 2
Myelopathy (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 4
Onychomycosis (Infections and infestations) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Colitis (Gastrointestinal disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Herpes zoster (Infections and infestations) | 3
Hydronephrosis (Renal and urinary disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Malaise (General disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Oral candidiasis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Tinea versicolour (Infections and infestations) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Arterial spasm (Vascular disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Candidiasis (Infections and infestations) | 1
Chalazion (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Herpes simplex (Infections and infestations) | 1
Hypertension (Vascular disorders) | 4
Influenza like illness (General disorders) | 1
Molluscum contagiosum (Infections and infestations) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tachycardia (Cardiac disorders) | 3
Traumatic renal injury (Injury, poisoning and procedural complications) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
BK virus infection (Infections and infestations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypocholesterolaemia (Metabolism and nutrition disorders) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Infected cyst (Infections and infestations) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 3
Overweight (Metabolism and nutrition disorders) | 1
Perinephric effusion (Renal and urinary disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Postoperative wound infection (Infections and infestations) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal vein thrombosis (Renal and urinary disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Staphylococcal infection (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
White blood cell count decreased (Investigations) | 2
Wound evisceration (Injury, poisoning and procedural complications) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Body tinea (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cerebral infarction (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Cyst (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Genital discharge (Reproductive system and breast disorders) | 1
Genital lesion (Reproductive system and breast disorders) | 1
Headache (Nervous system disorders) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Leukocyturia (Renal and urinary disorders) | 2
Liver function test abnormal (Investigations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Polycythaemia (Blood and lymphatic system disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Renal haemorrhage (Renal and urinary disorders) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 7
Amnesia (Nervous system disorders) | 1
Body temperature increased (Investigations) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Folliculitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Oedema (General disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Retinal haemorrhage (Eye disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Blood creatinine increased (Investigations) | 1
Depression (Psychiatric disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Incision site cellulitis (Infections and infestations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 3
Furuncle (Infections and infestations) | 2
Hiatus hernia (Gastrointestinal disorders) | 2
Influenza (Infections and infestations) | 4
Ischaemic ulcer (General disorders) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nocturia (Renal and urinary disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Tinea cruris (Infections and infestations) | 1
Troponin increased (Investigations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Urine output increased (Investigations) | 1
Vaginal infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.